CLINICAL TRIAL: NCT03653143
Title: Pilot Study of JASPER in Down Syndrome
Brief Title: JASPER Intervention in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nicole Baumer, Principle Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-P00025806
Record Dates: First submitted 2018-08-03; First posted 2018-08-31 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Down Syndrome, Trisomy 21
Keywords: Behavioral regulation; Emotional regulation; Social communication; Development
MeSH Terms: conditions — Down Syndrome; Emotional Regulation; Communication | interventions — Activator Appliances

STUDY DESIGN:
Intervention Model Description: Participants will initially undergo brief telephone screen to assess eligibility. Parents/guardians will complete surveys during the Baseline assessment and ERP/EEG testing will be done for participants who are able to undergo their assessments in-person. Participants will then be randomly assigned to either the treatment group or the control/waitlist group. The immediate group will start with 3 months of JASPER intervention and then have 3 months of their usual clinical care. The control/waitlist group will start with 3 months of their usual clinical care and then undergo 3 months of JASPER intervention. The 3-month treatment phase will involve weekly sessions with the JASPER interventionist, each 60 minutes long. Surveys and ERP/EEG assessments (as possible) will be repeated at the 3 month and at 6 month research visits for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Assessment #1 Baseline Visit >> 3 month JASPER intervention (weekly) >> Assessment #2 Research Visit >> 3 month treatment as usual >> Assessment #3 Research Visit
  Interventions: Behavioral: JASPER
- Control/Wait-list Group (Experimental): Assessment #1 Baseline Visit >> 3 month treatment as usual >> Assessment #2 Research Visit >> 3 month JASPER intervention >> Assessment #3 Research Visit
  Interventions: Behavioral: JASPER

INTERVENTIONS:
Behavioral: JASPER — JASPER is a therapist and parent-mediated intervention that (1) targets the foundations of social communication, (2) uses naturalistic behavioral strategies to increase the rate and complexity of social communication and (3) includes parents as implementers of the intervention to promote generalization across settings and to ensure maintenance. This intervention is individualized and centered around two key developmental domains critical for social communication function: joint engagement and joint attention.

SUMMARY:
The goal of this study is to determine whether JASPER (Joint Attention, Symbolic Play, Engagement, Regulation), which is an intensive, targeted early behavioral intervention focused on a developmentally based approach for teaching joint engagement, joint attention, and play skills can improve behavioral / emotional regulation, social communication skills, and developmental trajectories in Down syndrome (DS). The investigators will also explore the potential use of EEG and event-related potentials (ERP) as outcome measures, as this approach may help elucidate mechanisms of change in behavior and development, and may help explain differences in development of social communication skills in individuals with DS. EEG and ERP measure may also help to predict treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Trisomy 21
* Age 24-48 months
* Able to walk independently across a room
* Uses at least 5 words / signs
* English speaking
* Parent able to accompany participant to all study visits

Exclusion Criteria:

-Diagnosis of Mosaic / Translocation Down syndrome

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Joint Engagement | Administered at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  Joint engagement will be measured by coded videos of the Caregiver Child Interaction (CCX) session. CCX measures the amount of time that parent and child engage during a play session.

SECONDARY OUTCOMES:
Change in cognition | Administered at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  For in-person participation only, composite scores from the Mullen Scales of Early Learning (MSEL) will be used to measure cognition and language development. Composite scores are calculated averages based on MSEL subscales 1) Gross motor 2) Visual reception 3) Fine motor 4) Receptive language 5) Expressive language. Higher composite scores are associated with higher cognitive and language functioning.
Change in language, socialization, problem behavior, adaptive skills (part a) | Administered at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  Subscales of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) will be used to measure language, socialization, problem behaviors and adaptive skills. VABS-II subscales include 1) Communication 2) Daily living skills 3) Socialization, and 4) Motor skills. Behavior frequency is measured on a range of 0=Never to 1=Sometimes to 2=Usually.
Change in language, socialization, problem behavior, adaptive skills (part b) | Administered at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  The Aberrant Behavior Checklist-Community (ABC-C) will also be used to measure language, socialization, problem behavior, and adaptive skills for in-person participation. ABC-C subscales include 1) Irritability 2) Lethargy 3) Stereotypy 4) Hyperactivity, and 5) Inappropriate speech and are measured on a range of 0=not at all a problem to 3=the problem is severe in degree.
  The MacArthur-Bates Communicative Development Inventories (MB-CDI) will replace the ABC-C for virtual participation. The MB-CDI is a parent report instrument that captures important information about children's developing abilities in early language, including 1) Vocabulary comprehension 2) Production 3) Gestures, and 4) Grammar.
Change in social-communication skills (part a) | Administered at baseline assessment #1 (0 months) and assessment visit #3 (6 months)
  Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) will be used to measure social communication skills for in-person participation. ADOS-2 subscales include areas like 1) Language and communication and 2) Reciprocal social interaction. Items within each subscale are scored on unique ranges starting with 0=closest to mastery of behavior.
  The Autism Diagnostic Interview - Revised (ADI-R) will replace the ADOS for virtual participation. The ADI-R is a comprehensive parent interview that focuses on three functional domains of behavior that are not typically present in individuals without autism spectrum disorder. The three domains are: Language/Communication, Reciprocal Social Interactions, and Restricted, Repetitive, and Stereotyped Behaviors and Interests.
Change in social-communication skills (part b) | Administered at baseline assessment #1 (0 months) and assessment visit #3 (6 months)
  The Early Social Communication Scales (ESCS) is an experimental measurement that measures change in social-communication skills. It will be used for in-person participation only. The ESCS uses tasks to measure the frequency of initiation of and response to 1) Joint attention 2) Behavioral requests, and 3) Social interaction.
  The PICS will replace the ESCS for virtual participation. The PICS uses photographs to aid caregivers in understanding and identifying the specific behaviors of interest. Modeled after the ESCS, the PICS assesses various forms and functions of triadic attention in young children.
Change in joint attention skills | Administered at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  The Caregiver Child Interaction sessions (CCX) and Early Social Communication Scales (ESCS) or Pictorial Infant Communication Scale (PICS) will be used to measure changes in joint attention skills. ESCS, which will only be used for in-person participation, uses tasks to measure the frequency of the child's initiation and response (see above). The PICS will replace the ESCS for virtual participation. The PICS uses photographs to aid caregivers in understanding and identifying the specific behaviors of interest. Modeled after the ESCS, the PICS assesses various forms and functions of triadic attention in young children. The CCX, which will be used for in-person and virtual participation, measures the amount of time that parent and child engage during a play session.
Change in play levels | Administered at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  Flexibility and diversity of play will be coded from the Structured Play Assessment (SPA) for in-person participation only. Different toys are presented to the child, and play interaction is measured in terms of 1) Functional play types 2) Symbolic play types, and 3) Play level.

OTHER OUTCOMES:
Change in social-communication skills (in relation to electrophysiology) | EEG will be measured at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  Resting state electroencephalogram (EEG) power will be measured as a potential moderator of treatment on change in joint engagement (baseline to end of treatment). EEG procedures will be conducted using a previously established JASPER EEG protocol.
Change in social-communication skills (in relation to electrophysiology) | ERP visual, auditory, and face processing will be measured at baseline assessment #1 (0 months), assessment visit #2 (3 months), and assessment visit #3 (6 months)
  Electroencephalogram (EEG) is brain monitoring method that will be used to measure brain activity. EEG power will first be measured during "resting state". Brain activity in response to low-level visual processing, low-level auditory processing, and face processing will then be measured using event-related potentials (ERPs).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Baumer, MD, MEd, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Kasari C, Gulsrud A, Freeman S, Paparella T, Hellemann G. Longitudinal follow-up of children with autism receiving targeted interventions on joint attention and play. J Am Acad Child Adolesc Psychiatry. 2012 May;51(5):487-95. doi: 10.1016/j.jaac.2012.02.019. Epub 2012 Apr 6. PMID 22525955